CLINICAL TRIAL: NCT00514618
Title: Outpatient Cervical Ripening and Labor Induction With Orally Administered Misoprostol for Term Pregnancies Complicated by Diabetes Mellitus
Brief Title: Outpatient Cervical Ripening With Orally Administered Misoprostol in Diabetics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: MemorialCare Health System (Other)
Collaborators: Long Beach Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 334-06 [no UCI HS#]
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2023-10-23 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-09

CONDITIONS: Diabetes, Gestational
Keywords: Term Pregnancy; Diabetes; Cervical Ripening; Induction; misoprostol; Term Gestational Diabetics
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): patients will be treated with misoprostol 50 mcg PO
  Interventions: Drug: Misoprostol
- 2 (Placebo Comparator): patients will receive placebo (Vitamin C)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Misoprostol — patients will be treated with misoprostol 50 mcg PO q day for two days (days 1 and 4)
  Other Names: Cytotec
  Arms: 1
Dietary Supplement: Placebo — patients will receive placebo (vitamin C) q day for two days (days 1 and 4)
  Arms: 2

SUMMARY:
A. Null Hypothesis:

In term pregnancies complicated by diabetes, there is no difference in the time interval from start of induction to delivery when outpatient cervical ripening and labor induction is initiated with orally administered misoprostol, a prostaglandin El analogue, compared to placebo.

B. Specific aims:

1. Demonstrate that oral misoprostol is effective for cervical ripening compared to placebo when given in an outpatient basis to women with pregnancies complicated by diabetes mellitus.
2. Demonstrate that oral misoprostol can be administered safely in an outpatient setting. The patients will be observed for a period of four hours in an outpatient antepartum testing unit after the medication is administered to demonstrate fetal well being and verify that there is no evidence of uterine hyperstimulation. (We acknowledge that markers of serious adverse maternal and neonatal outcomes are rare, and can only be adequately addressed in large multicenter trials.)
3. Assess the cost differential in inpatient and outpatient utilization of misoprostol for cervical ripening and labor induction. In order to estimate the impact that outpatient cervical ripening may have on total hospitalization costs, we will use daily hospital charges and published data regarding pharmaceutical costs.

DETAILED DESCRIPTION:
The study proposed is a single center study. Study participants will be recruited from the high risk obstetrical diabetic resident clinic, the Magella Women's Perinatal Group, and Fetal Diagnostics at Miller Children's hospital. The resident clinic is supervised by the faculty from the division of Maternal Fetal Medicine from the department of Obstetrics and Gynecology. Patients with class A1, A2 diabetes mellitus at term who are usually considered for inpatient cervical ripening and labor induction will be approached for participation in the study. Informed consent will be obtained by members of the perinatal research team.

One hundred twenty-eight patients will be enrolled to assess treatment efficacy. Sixty four patients will be treated with misoprostol 50mcg PO q day for two days (days 1 and 4) and sixty four patients will receive placebo (vitamin C) q day for two days (days 1 and 4) for cervical ripening and labor induction.

Sample size calculations were performed assuming that 50% of untreated patients will deliver within 7 days of entry. Using an estimate that a 50% increase in this number to 75% would be clinically important, and assuming a Type I error of 0.05 and a Type II error of 0.2, we calculated that a sample size of 58 patients in each group was necessary. The test was one-sided. Assuming a 10% loss to follow-up rate, sixty four patients will be needed in each group.

A predetermined randomization schedule for the 128 patients has been established and the randomization assignments placed in opaque, sealed envelopes. The randomization was performed using a computer-generated random number table. The pharmacy will prepare and distribute the study medication according to the randomization schedule after eligible participants sign the informed consent. Once a patient is randomized, the pharmacy will be contacted to provide the medications to the research/antepartum testing unit nurse.

The proposed study length is two years, or the time needed to enroll 128 total participants. Each individual's total participation time is that needed to complete the protocol. After delivery, the prenatal and hospital charts of each participant will be reviewed and data abstracted.

Outpatient Procedures:

1. Initial complete history and physical exam by physicians in the clinics, including cervical exam.
2. The patients will be sent to the antepartum testing unit to undergo a non-stress test and amniotic fluid index measurement as indicators of fetal well-being.
3. Candidates will be approached for study participation and informed consent obtained.
4. The pharmacy will be contacted for randomization and provision of the study medications.
5. A research nurse or physician, trained in labor and delivery, will be responsible for administration of the study medication (50 mcg misoprostol or placebo).
6. The patient will be observed in the antepartum testing unit for a period of 4 hours after receipt of the study medication.

   1. Adequate uterine activity will be defined as >=3 uterine contractions (UC's) in 10 minutes. Inadequate uterine activity will be defined as <=2/10 minutes. Continued adequate uterine activity will require continued observation on the labor and delivery unit. If there is cessation of uterine activity while under observation on labor and delivery and the fetal heart rate pattern remains reassuring, the patient will be discharged home to return in three to four days for a second dose of medication or oxytocin, as appropriate.
   2. Adequate cervical ripening: If, following receipt of the medication, a patient demonstrates a change in cervical score to >6, she will be admitted for delivery.
   3. If spontaneous labor ensues, or the patient demonstrates uterine hyperstimulation, she will be transferred to the labor and delivery unit.
7. If after the period of observation, the fetal heart rate testing remains reassuring and the patient is not in labor or developed an adequate contraction pattern, she will be discharged home.
8. If discharged home, the patient will be instructed to return 3 or 4 days later (coincident with standard antepartum testing protocol) for re-evaluation for a second dose of the study medication.
9. On the second day coincident with antepartum testing, a repeat cervical examination will be performed by a research nurse, resident or attendant physician. Non Stress Test will be performed. If the Bishop score is >6, the patient will be admitted to labor and delivery for oxytocin augmentation of her labor. If the Bishop score is less than this, the Non Stress Test is reactive, amniotic fluid index normal, and uterine activity is minimal, she will be administered a second dose of 50 mcg of oral misoprostol. Observation in the antepartum testing unit will be for 4 hours. Again, if labor does not ensue and the fetal heart rate remains reassuring, the patient will be sent home again with instructions to return 3-4 days later coincident with standard NST.
10. On the morning of the seventh day (one week after enrollment and receipt of first dose of oral misoprostol, 39 ½ weeks' gestational age), the patient will be admitted to the labor and delivery unit to undergo inpatient cervical ripening with oral misoprostol, or oxytocin induction or augmentation as appropriate.
11. All patients who are discharged home on days 1 and 4 will be instructed to observe for signs of labor or ruptured membranes, and to assess fetal movement while at home. They will be instructed to return to the emergency room if they experience uterine contractions occur as often as every 5 minutes for 1 hour, rupture of membranes, heavy vaginal bleeding or decreased fetal movement.
12. A 24-hour emergency phone number will be provided for all patients enrolled into this study protocol.
13. Labor management during the active phase of labor on the unit will be at discretion of the managing physician.

Labor and delivery admission procedure:

1. Intravenous access will be obtained.
2. Standard laboratory studies will be drawn, including Type and screen, complete blood count, capillary blood glucose.
3. Continuous external fetal monitoring and external tocodynamometry will be utilized.
4. A cervical examination will be performed by the physician.

NOTE: These (1-4) are the standard procedures applied to patients admitted to labor and delivery.

Misoprostol Inpatient Administration:

Those patients who remain with an unripened cervix and with uterine contractions less than 12/hour after completion of days 1 and 4 of outpatient treatment will be candidates to receive misoprostol as an inpatient on day 7 per the following protocol.

1. The dosing schedule will be as follows: 100 micrograms of misoprostol given orally every 4 hours to a maximum of 6 doses. (The medication will be provided by the pharmacy).

   A. The maximum cervical ripening period will be 24 hours. After 24 hours of misoprostol, if the patient has not entered active labor, the induction process may be continued with oxytocin as necessary.

   B. Continued, regular uterine activity (3 uterine contractions in a 10 minute period) will preclude repeat dosing.
2. In the event of spontaneous rupture of membranes, the patient will receive no further doses of misoprostol. Oxytocin may be utilized to augment labor at the discretion of managing physician.
3. If the patient develops a uterine contraction abnormality as defined below, either terbutaline, 0.25 mg IV or SQ or MgSO4 intravenous infusion may be administered as necessary. If such abnormalities are encountered during oxytocin administration, the infusion will be discontinued and the same treatment may be utilized.
4. The maximum time period for cervical ripening with misoprostol is 24 hours, which may be followed immediately by an adequate trial of oxytocin, which usually will not exceed 24 hours. Thus, no inpatient cervical ripening/induction attempt will exceed 48 hours.

Oxytocin Induction/ Augmentation (as necessary):

1) These patients will receive oxytocin infusions according to the standard labor and delivery protocol at Miller and Children's Hospital.

Study Outcomes:

The primary outcome measure will be the time interval from start of induction to delivery. Other outcome measures will be number of doses of medication required, oxytocin requirements, and route of delivery. The number of patients admitted to labor and delivery in active labor will also be assessed as will interval changes in Bishop's score after application of medication. Also intrapartum complications including uterine hyperstimulation, fetal distress and excessive bleeding at the time of delivery will be compared, as will adverse maternal and neonatal outcomes, e.g., development of endometritis or admission to the NICU respectively.

Expected Outcomes:

We anticipate that approximately 20% of patients after receiving misoprostol will enter the active phase of labor and require transfer to labor and delivery. We also anticipate that we will find significant differences in Bishop's scores between the two groups from day 1 and 4, and find significantly shorter time intervals from start of induction to delivery in those patients who receive the active agent.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation
2. Intact membranes
3. Bishop score <= 4
4. Uterine contractions <=12/hour
5. Cephalic presentation
6. Estimated gestational age of at least 38 weeks by ACOG dates
7. An amniotic fluid index (AFI) >5 cm
8. Reactive Non Stress Test
9. Class A1, A2 diabetes
10. Good compliance with clinic visits and home glucose monitoring

Exclusion Criteria:

I. Fetal Factors

1. Multiple Gestation
2. Presence of fetal distress/non-reassuring FHR pattern
3. Malpresentation, including breech
4. EFW > 4500 gm or other evidence of cephalo-pelvic disproportion
5. EFW < 2000 gm

II. Maternal Factors

1. Frequent uterine contractions >= 12/hour
2. Ruptured membranes
3. Placenta previa or unexplained vaginal bleeding
4. Vasa previa
5. Active herpes simplex
6. Glaucoma or elevated intraocular pressure
7. Renal or hepatic dysfunction
8. Previous Cesarean delivery or history of uterine surgery
9. Evidence of chorioamnionitis or maternal fetal >= 100.4 degrees F
10. Significant cardiac lesion or cardiovascular disease
11. Severe asthma
12. Parity >=6

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Wing, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI has left the institution. Efforts were exhausted in attempting to contact the PI/study team members. No study data are available
Pre-assignment Details: The PI has left the institution. Efforts were exhausted in attempting to contact the PI/study team members. No study data are available.
Groups:
- 1 - Misoprostol Treated: patients will be treated with misoprostol 50 mcg PO
- 2 - Placebo: patients will receive placebo (Vitamin C)
Period: Overall Study
Arm/Group | 1 - Misoprostol Treated | 2 - Placebo
Started (The PI has left the institution. Efforts were exhausted in attempting to contact the PI/study team members. No study data are available. No UCI protocol.) | 5 | 0
Completed (The PI has left the institution. Efforts were exhausted in attempting to contact the PI/study team members. No study data are available. No UCI protocol.) | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data was collected.
Groups:
- 1 - Misoprostol Treated: patients will be treated with misoprostol 50 mcg PO
  Misoprostol: patients will be treated with misoprostol 50 mcg PO q day for two days (days 1 and 4)
- 2 - Placebo: patients will receive placebo (Vitamin C)
  Placebo: patients will receive placebo (vitamin C) q day for two days (days 1 and 4)
- Total: Total of all reporting groups
Arm/Group | 1 - Misoprostol Treated | 2 - Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be the Time Interval From Start of Induction to Delivery.
Description: Demonstrate that oral misoprostol is effective for cervical ripening compared to placebo when given in an outpatient basis to women with pregnancies complicated by diabetes mellitus.
  The study was terminated, and no study data and/or analyzed. No study data are available.
Time Frame: induction to delivery
Population: No data was collected.
Groups:
- 1 Misoprostol 50mcg: patients will be treated with misoprostol 50 mcg PO
- 2 Placebo: patients will receive placebo (Vitamin C)
Arm/Group | 1 Misoprostol 50mcg | 2 Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Demonstrate That Oral Misoprostol Can be Administered Safely in an Outpatient Setting.
Description: The study was terminated, and no study data and/or analyzed. No study data are available.
Time Frame: The PI has left the institution. Efforts were exhausted in attempting to contact the PI/study team members. No study data are available.
Population: No data was collected.
Arm/Group | 1 Misoprostol 50mcg | 2 Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Other Outcome Measures Will be Number of Doses of Medication Required, Oxytocin Requirements, and Route of Delivery.
Description: No data was collected.
Time Frame: induction to delivery
Population: No data was collected.
Arm/Group | 1 Misoprostol 50mcg | 2 Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious Adverse Events and/or Other Adverse Events data were not collected.
Description: No data was collected.
Arm/Group | 1 - Misoprostol Treated | 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 - Misoprostol Treated (N=0) | 2 - Placebo (N=0)
No adverse events were collected (Pregnancy, puerperium and perinatal conditions) | 0 | NA — There were no serious adverse events information collected.

LIMITATIONS AND CAVEATS:
No data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No